CLINICAL TRIAL: NCT04463797
Title: Effects of Square-stepping Exercise on Frailty and Cognitive Function in Elderly With Frailty and MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM109044F
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2022-09

CONDITIONS: Frailty; Mild Cognitive Impairment
Keywords: Frailty; Mild cognitive impairment; Square-stepping exercise; Cognitive function
MeSH Terms: conditions — Frailty; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Square-stepping exercise group (Experimental): Square-stepping exercise
  Interventions: Other: Square-stepping exercise
- Control group (Active Comparator): Whole-body stretching and upper extremity strengthening
  Interventions: Other: Stretching and strengthening

INTERVENTIONS:
Other: Square-stepping exercise — The square-stepping exercise is a low-cost indoor program to improve lower extremities fitness and cognitive function.
  Arms: Square-stepping exercise group
Other: Stretching and strengthening — whole-body stretching and upper extremity strengthening
  Arms: Control group

SUMMARY:
This is a single-blinded, randomized controlled trail with pre- and post-measurements. The inclusion criteria are: (1) age between 65 to 90 years old, (2) the presence of at least one of the 5 physical characteristics defined by Fried, (3) with mini-mental state examination (MMSE) score≧24 and Montreal cognitive assessment (MoCA) score < 26, and (4) ability to walk independently for 1 min without assistive devices. The exclusion criteria are: unstable physical condition, any neurological, psychiatric disorder, or diagnosed with learning disability which may affect participation in this study. Twenty-eight elderly will be recruited, and randomly assigned to one of two groups: square-stepping exercise (SSE) group (n=14) or control group (n=14). The intervention for both group will be 50 minutes per session, 3 sessions per week for 8 weeks. The primary outcomes include frailty status indicated by Fried frailty criteria, and global cognitive function indicated by MoCA score. Secondary outcomes include frailty and MCI reverse rate, attention and memory, executive function, physical performance, and brain activation.

DETAILED DESCRIPTION:
Background and purpose:

Frailty is a continuous decline of multiple physiological systems along with aging. Common characteristics of frailty are fatigue, weakness, weight loss, slowness, and low physical activity. Brain changes accompanying frailty may lead to cognitive decline. Moreover, evidence showed positive relations between frailty and cognitive decline. Frailty with cognitive decline increases the risk of various adverse outcomes, such as disability, hospitalization, incidence of dementia, loss of daily activity functioning, and poor quality of life. Physical exercise training is a common intervention for frail elderly; however, most studies applying physical exercise to frail elderly are for enhancing physical performance, few are for improving cognitive function. On the other hand, the square-stepping exercise has been proven to be beneficial to healthy older adults for both physical performance and cognitive function, but it's application for frail elderly is scarce. Therefore, the purpose of this study is to explore the effects of the square-stepping exercise on frailty and cognitive function in elderly with frailty and mild cognitive impairment (MCI).

Method:

This is a single-blinded, randomized controlled trail with pre- and post-measurements. The inclusion criteria are: (1) age between 65 to 90 years old, (2) the presence of at least one of the 5 physical characteristics defined by Fried, (3) with mini-mental state examination (MMSE) score≧24 and Montreal cognitive assessment (MoCA) score < 26, and (4) ability to walk independently for 1 min without assistive devices. The exclusion criteria are: unstable physical condition, any neurological, psychiatric disorder, or diagnosed with learning disability which may affect participation in this study. Twenty-eight elderly will be recruited, and randomly assigned to one of two groups: square-stepping exercise (SSE) group (n=14) or control group (n=14). The intervention for both group will be 50 minutes per session, 3 sessions per week for 8 weeks. The primary outcomes include frailty status indicated by Fried frailty criteria, and global cognitive function indicated by MoCA score. Secondary outcomes include frailty and MCI reverse rate, attention and memory, executive function, physical performance, and brain activation.

SPSS 25.0 will be used for data analysis, with significant level set at 0.05. Repeated measures two-way analysis of variance (ANOVA) with Tukey's post-hoc analysis will be used to compare between time (pre-test, post-test) and between groups. Chi-square test (χ2 test) will be applied comparing data of frailty/ MCI reverse rate.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 to 90 years old
* Presence of at least one of the 5 physical characteristics of frailty defined by Fried
* Mini-mental state examination (MMSE) score more than or equal to 24
* Montreal cognitive assessment (MoCA) score less than 26
* Ability to walk independently for 1 min without assistive devices

Exclusion Criteria:

* Unstable physical condition
* Any neurological or psychiatric disorder
* Diagnosed with learning disability which may affect participation in this study

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Fried frailty criteria | 10 minutes
  To assess the frailty status, score ranges from 1 to 5.
The Montreal Cognitive Assessment | 8 minutes
  Evaluating global cognitive function, score ranges from 1 to 30.

SECONDARY OUTCOMES:
Frailty reverse rate | 2 minutes
  The percentage of subjects in each group who reverse from prefrail to robust, and frail to prefrail or robust.
MCI reverse rate | 2 minutes
  The percentage of subjects in each group who reverse from MCI to normal cognitive function.
Digit Span Test | 8 minutes
  Attention and memory
Trail Making Test | 8 minutes
  Executive function
Timed Up and Go Test | 5 minutes
  Dynamic balance and mobility
6-minute walk test | 10 minutes
  Endurance and physical fitness
Lower extremity strength | 5 minutes
  Measuring lower extremity strength of the subject with a dynamometer.
Brain activation | 30 minutes
  Measured by a wearable functional near-infrared spectroscopy system in bilateral prefrontal cortex (PFC), premotor cortex (PMC), supplementary motor area (SMA).

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided